CLINICAL TRIAL: NCT05768672
Title: Investigating the Relationship Between the Sense of Smell and Cognitive Inhibition in Obesity: a Behavioural Experiment.
Brief Title: The Sense of Small and Inhibition in Obesity
Acronym: Smell_OB
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Università degli Studi di Trento (Other)
Responsible Party: Sponsor
Other Study IDs: 21C221
Record Dates: First submitted 2023-02-22; First posted 2023-03-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: obesity; smell; food; cognitive inhibition
MeSH Terms: conditions — Obesity; Anosmia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Right-handed Individuals diagnosed with obesity will be recruited at the beginning of a rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy).
  Interventions: Behavioral: Experimental Task
- Controls: Age-matched, right-handed, individuals with a healthy weight recruited outside the hospital through personal contacts of the researchers and word-of-mouth
  Interventions: Behavioral: Experimental Task

INTERVENTIONS:
Behavioral: Experimental Task — The main task is an olfactory version of a traditional Go/No-Go task (Albayay et al., 2019): it includes the delivery of either an odour or clean air prior to the presentation of a visual target Moreover, all participants will be assessed with the italian version of the Stroop color and word test (Caffarra et al., 2004) to evaluate inhibition, together with selective and sustained attention. This neuropsychological test consists of three tables, showing color words (W), colored circles (C), and color words printed in incongruent ink (i.e., red printed in blue ink, CW), respectively. The Stroop effect consists of a delayed response when words have to be named according to the color of the ink, ignoring the meaning of the printed word.

SUMMARY:
The aim of this research is to verify whether inhibitory control ability is different between a group of individuals with obesity and a group of individuals with normal weight in the presence of olfactory stimuli, different for valence, edibility (food versus no-food), and caloric density (high-calorie vs low-calorie content) of foods associated with odours.

ELIGIBILITY:
Inclusion criteria:

* Right-handed
* diagnosis of obesity (i.e., the level of body mass index (BMI) higher or equal to 30).

Exclusion criteria:

* Concurrent neurological, neurodevelopmental (e.g., autism), motor, somatosensory and/or psychiatric disorders.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with obesity will be recruited at the beginning of a rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Error % | baseline
  Percentage of the invalid answers, meaning when the participant erroneously press the key (i.e., answer) in the no-go (invalid) trials. This represents an index of inhibitory difficulty in the experimental task. This score will be computed according to Albayay and colleagues (2019).

SECONDARY OUTCOMES:
Interference Error | baseline
  It will computed according to the following formula:
  score = CW - ((W + C)/2). The lower is the score, the best is the performance. Notably for each condition (W, C, and CW) the number of error can range from O (no error) to 36 (maximun number of error). This computation derives from the seminal article for the Italian version of the test (Caffarra et al., 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Tagini, PhD, Principal Investigator — IRCCS Istituto Auxologico Italiano
Locations (1):
- IRCCS Istituto Auxologico Italiano - Ospedale San Giuseppe, Piancavallo, VCO, Italy